CLINICAL TRIAL: NCT05343832
Title: Detection Evaluation of a Novel Blood-based DNA Methylation Assay in Early-stage Hepatocellular Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Genetron Health (Industry)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou eighth People's Hospital ,Guangzhou Medilcal University (Unknown); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); West China Hospital (Other); Beijing Youan Hospital,Capital Medical University Beijing Institute of Hepatology (Unknown); Ruijin Hospital (Other); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Wuxi No.5 People's Hospital (Unknown); Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20210280
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trail is a multi-center,prospective observational study aimed to detect early-stage Hepatocellular Carcinoma by a Novel Blood-based DNA Methylation Assay(named Genetron HCC Methylation PCR Kit ). The accuracy of the kit will also be evaluated . The trail will be enroll approximately 4816 participants, including participants with HCC or benign diseases, and high risk factors for liver cancer.

DETAILED DESCRIPTION:
Diagnostic performance evaluation:

Alpha-fetoprotein (AFP), liver ultrasound (US), dynamic contrast enhanced MRI and the kit examination will be performed on high-risk participants of primary liver cancer.

For subjects with typical imaging findings of hepatocellular carcinoma but an intrahepatic nodule diameter of ≤2 cm, an imaging study will be added to the above.

According to the clinical diagnostic criteria of primary liver cancer, the diagnostic performance of the kit, liver ultrasound examination (US) combined with alpha fetoprotein (AFP) detection will be evaluated, and the sensitivity of the kit, the kit combined with AFP, the kit combined with AFP and US, AFP combined with US screening for primary liver cancer will be compared.

Test performance evaluation:

Plasma samples of patients with and without HCC diagnosed according to the clinical diagnostic criteria of primary HCC will be collected and examined simultaneously by the kit and high-throughput human methylation sequencing (NGS sequencing).

ELIGIBILITY:
Diagnostic performance evaluation:

Inclusion Criteria:

1. Have high risk factors for liver cancer such as HBV and/or HCV infection, alcoholic liver disease, non-alcoholic steatohepatitis, long-term consumption of food contaminated with aflatoxin, liver cirrhosis caused by various other reasons, and family history of liver cancer Wait;
2. I or my legal representative can read, understand and sign the informed consent;
3. Agree to provide blood samples, be able to receive imaging examinations and have good clinical compliance;
4. The complete clinical basic information includes: the patient's unique traceability number (ID number/outpatient clinic number/medical insurance card number), age, gender, etc.

Exclusion Criteria:

1. pregnant women;
2. Have received an organ transplant;
3. Diagnosed with other tumors;
4. The investigators judged that they were not eligible for inclusion.

Test performance evaluation:

Inclusion Criteria:

1. Confirmed primary hepatocellular carcinoma or confirmed non-HCC;
2. I or my legal representative can read, understand and sign the informed consent;
3. Agree to provide blood samples and have good clinical compliance;
4. The basic clinical information is complete, including: the patient's unique traceability number (ID number/outpatient clinic number/medical insurance card number), age, gender, imaging and/or pathological diagnosis results (for patients with primary liver cancer), imaging examination confirmed non-identical Liver cancer (non-HCC patients).

Exclusion Criteria:

1. pregnant women;
2. Have received an organ transplant;
3. Non-HCC patients diagnosed with other tumors;
4. Patients with primary hepatocellular carcinoma combined with other tumors;
5. The investigator judges that they are not eligible for inclusion.

Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with primary hepatocellular carcinoma, or with high risk factors for liver cancer such as HBV and/or HCV infection, alcoholic liver disease, non-alcoholic steatohepatitis, long-term consumption of food contaminated with aflatoxin, various other causes of liver cirrhosis, and patients with a family history of liver cancer, etc.
Sampling Method: Non-Probability Sample
Enrollment: 4816 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-03-05 (Estimated); Study Completion 2023-04-25 (Estimated)

PRIMARY OUTCOMES:
All plasma samples and imaging results will be used to evaluate diagnostic(sensitivity and specificity) of the kit. | 2 months
  Alpha-fetoprotein (AFP), liver ultrasound (US), dynamic contrast enhanced MRI and the kit examination will be performed on high-risk participants of primary liver cancer.
  For subjects with typical imaging findings of hepatocellular carcinoma but an intrahepatic nodule diameter of ≤2 cm, an imaging study will be added to the above.
  According to the clinical diagnostic criteria of primary liver cancer, the diagnostic performance of the kit, liver ultrasound examination (US) combined with alpha fetoprotein (AFP) detection will be evaluated, and the sensitivity of the kit, the kit combined with AFP, the kit combined with AFP and US, AFP combined with US screening for primary liver cancer will be compared.
Plasma samples of patients with and without HCC to evaluate test performance(accuracy) of the kit. diagnostic(sensitivity and specificity) of the kit. | 2 months
  Following the principle of simultaneous blinding, blood samples were collected from liver cancer patients and non-HCC patients who had been diagnosed according to the clinical diagnostic criteria for primary liver cancer. The subjects were coded, and the selected samples were tested by the kit and the comparison method high-throughput human methylation sequencing (NGS sequencing method), and the test results were compared.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Beijing Youan Hospital,Capital Medical University Beijing Institute of Hepatology, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China School of Medicine/West China Hospital of Sichuan University, Chengdu
  - Guangzhou eighth People's Hospital ,Guangzhou Medilcal University, Guangzhou
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Nantong Tumor Hospital, Nantong
  - Ruijin Hospital, Shanghai Jiaotong University School, Shanghai
  - Wuxi No.5 People's Hospital, Wuxi
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT05343832/Prot_000.pdf